CLINICAL TRIAL: NCT05934188
Title: Role of the Gut-microbiota on Ageing and Neurodegeneration: a Clinical and Brain Imaging Study
Brief Title: Exploring the Gut-Brain Axis in Ageing and Neurodegeneration
Acronym: GutBrain
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Collaborators: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other); Università Ca' Foscari Venezia (Unknown)
Responsible Party: Principal Investigator, Nicola Filippini, Principal Investigator, IRCCS San Camillo, Venezia, Italy
Other Study IDs: 2022.13; RF-2021-12372224 (Other Grant/Funding Number: Ministry of Health)
Record Dates: First submitted 2023-06-09; First posted 2023-07-06 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Healthy; Prodromal Alzheimer's Disease; Parkinson Disease; Multiple Sclerosis
Keywords: MRI; Microbiota; Stool sample; Blood sample; Neuropsychological assessment; Neuroimaging; Biomarkers for brain disorders
MeSH Terms: conditions — Parkinson Disease; Multiple Sclerosis | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Young Healthy Subjects (N = 40): * 20-50 years old
  * Cognitively healthy (Mini-Mental State examination ≥ 26)
  * Absence of significant neurological disorders
  Interventions: Diagnostic Test: Magnetic Resonance Imaging; Behavioral: Neuropsychological protocol; Behavioral: Eating habits; Diagnostic Test: Microbiome analyses; Diagnostic Test: Inflammatory markers
- Old Healthy Subjects (N = 40): * 60-90 years old
  * Cognitively healthy (Mini-Mental State examination ≥ 26)
  * Absence of significant neurological disorders
  Interventions: Diagnostic Test: Magnetic Resonance Imaging; Behavioral: Neuropsychological protocol; Behavioral: Eating habits; Diagnostic Test: Microbiome analyses; Diagnostic Test: Inflammatory markers
- Patients with prodromal Alzheimer's Disease (N = 40): * Subjective cognitive complaint (corroborated by the informant)
  * Episodic memory deficit on neuropsychological testing
  * Clinical Dementia Rating = 0.5
  * Mini-Mental State Examination (MMSE) > 23
  * Independently functioning in activities of daily living
  Interventions: Diagnostic Test: Magnetic Resonance Imaging; Behavioral: Neuropsychological protocol; Behavioral: Eating habits; Diagnostic Test: Microbiome analyses; Diagnostic Test: Inflammatory markers; Diagnostic Test: Alzheimer's Disease biomarkers
- Patients with Parkinson's Disease (N = 40): * Recent diagnosis of Parkinson's Disease
  * Mild-moderate score at the Unified Parkinson's Disease Rating Scale (UPDRS)
  * Cognitively healthy (Mini-Mental State examination ≥ 26)
  * In case of taking medications for Parkinson's Disease: stable dosage for at least 6 months
  Interventions: Diagnostic Test: Magnetic Resonance Imaging; Behavioral: Neuropsychological protocol; Behavioral: Eating habits; Diagnostic Test: Microbiome analyses; Diagnostic Test: Inflammatory markers
- Patients with Multiple Sclerosis (N = 40): * Recent diagnosis of relapsing-remitting Multiple Sclerosis
  * Expanded Disability Status Scale score ≤ 4.0
  * Cognitively healthy (Mini-Mental State examination ≥ 26)
  * In case of taking medications for Multiple Sclerosis: stable dosage for at least 6 months
  Interventions: Diagnostic Test: Magnetic Resonance Imaging; Behavioral: Neuropsychological protocol; Behavioral: Eating habits; Diagnostic Test: Microbiome analyses; Diagnostic Test: Inflammatory markers

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging — The Magnetic Resonance Imaging protocol will comprise both structural and functional sequences.
Behavioral: Neuropsychological protocol — Neuropsychological tests will be administered to participants to assess general cognitive state and a range of high-level cognitive functions (memory, executive, language). In addition, disease-specific tests will be administered to patients to investigate disease staging and the level of disability and autonomy.
Behavioral: Eating habits — Information on eating habits will be derived from food questionnaires.
Diagnostic Test: Microbiome analyses — The Microbiome analyses will be derived from a stool sample (16S rRNA sequencing targeted metagenomic analyses).
Diagnostic Test: Inflammatory markers — Inflammatory markers will be evaluated in terms RNA expression level in plasma blood sample.
Diagnostic Test: Alzheimer's Disease biomarkers — The Alzheimer's Disease biomarkers will be measured in the plasma of prodromal Alzheimer's Disease patients.
  Groups: Patients with prodromal Alzheimer's Disease (N = 40)

SUMMARY:
Neurodegenerative diseases are a major health concern due to their growing societal implications and economic costs. The identification of early markers of pathogenic mechanisms is one of the current main challenges. The gut-brain axis has become a primary target because of its transversal role across the neurodegenerative spectrum and its effect on cognition. However, despite recent progress, how changes in the gut-microbiota composition can affect the human brain is still unclear.

The goal of this observational study is to characterise the gut-microbiota composition associated with alterations in brain structure and function during the ageing process and across neurodegenerative disorders. This is based on recent studies showing that changes in the human brain and in the microbiota composition, can indicate very sensitively and in a predictive way pathological development and, consequently, be used as markers of neurodegenerative diseases.

The main questions it aims to answer are:

* How variation in the gut-microbiota composition correlates with the normal brain ageing trajectory?
* How dysregulation in the gut-microbiota correlates with pathological changes in brain regions in specific neurodegenerative disorders?
* Can the impact of the gut-microbiota on the brain be modulated by blood biomarkers?

The investigators will recruit 40 young healthy participants, 40 old healthy participants, 40 participants with prodromal Alzheimer's Disease, 40 participants with Parkinson's Disease and 40 participants with Multiple Sclerosis.

Participants will undergo the following examinations:

* Magnetic Resonance Imaging
* Analysis of a stool sample
* Analysis of a blood sample
* Neuropsychological assessment
* Questionnaires on eating habits

DETAILED DESCRIPTION:
Recent studies show that alterations in the microbiota profile has been observed in the ageing process and across neurodegenerative disorders and it has been associated with cognitive decline and disease-specific clinical symptoms.

The objective of this multicenter observational cross-sectional cohort study is to characterise how changes in the gut-microbiota profile may affect brain changes during the physiological ageing processes and across neurodegenerative disorders with different etiopathogenesis.

The investigators will combine novel magnetic resonance imaging and biological techniques to test these hypotheses:

1. Specific functional and structural changes, which reflect unsuccessful compensatory mechanisms to counteract ageing, are associated with changes in the gut-microbiota composition.
2. Neurodegenerative disorders (prodromal Alzheimer's Disease, Parkinson's Disease, Multiple Sclerosis) show unique changes in the gut-microbiome profile, associated with specific structural and functional brain changes.
3. The microbiota profile characterizing the unsuccessful ageing and different neurodegenerative diseases is associated with alterations in blood biomarkers.

For this study the investigators plan to recruit 80 healthy subjects divided into two groups (40 subjects aged 20-50 years and 40 subjects aged 60-90 years) and 120 patients divided into three groups (40 patients with prodromal Alzheimer's Disease, 40 patients with Parkinson's Disease and 40 patients with Multiple Sclerosis).

All participants will undergo a multimodal Magnetic Resonance Imaging protocol to study the brain structure and function and a detailed neuropsychological protocol to assess cognitive functioning. In addition, stool and blood samples will be collected to investigate the gut-microbiota composition and the presence of inflammatory markers, respectively. Participants will also be asked to fill out questionnaires on eating habits.

There are no known risks or long-term side effects related to Magnetic Resonance Imaging. The performance of the examination does not involve physical or mental impairment.

The study does not directly benefit the participant. However, participation in the study will increase knowledge in the area of the relationship between the gut microbiota and the brain, providing potential new knowledge useful for preventing the risk of developing neurodegenerative processes.

The study takes place at San Camillo IRCCS S.r.l. (70 Alberoni street, Lido VE, 30126, Italy IT).

The study started on 01/05/2023 and the end is planned for 30/04/2026. The submitted study is funded by the Ministry of Health through a finalized research call won by Principal Investigator, Dr. Nicola Filippini, and approved by Ethics Committee for Clinical Trials of the Province of Venice and IRCCS San Camillo, Azienda ULSS 3 Serenissima.

ELIGIBILITY:
INCLUSION CRITERIA:

Healthy Young and Old Subjects:

* 20-50 or 60-90 years old
* Cognitively healthy (Mini-Mental State examination ≥ 26)
* Absence of significant neurological disorders

Patients with prodromal Alzheimer's Disease:

* Subjective cognitive complaint (corroborated by the informant)
* Episodic memory deficit on neuropsychological testing
* Clinical Dementia Rating = 0.5
* Mini-Mental State Examination (MMSE) > 23
* Independently functioning in activities of daily living

Patients with Parkinson's Disease:

* Recent diagnosis of Parkinson's Disease
* Mild-moderate score at the Unified Parkinson's Disease Rating Scale (UPDRS)
* Cognitively healthy (Mini-Mental State examination ≥ 26)
* In case of taking medications for Parkinson's Disease: stable dosage for at least 6 months

Patients with Multiple Sclerosis:

* Recent diagnosis of relapsing-remitting Multiple Sclerosis
* Expanded Disability Status Scale score ≤ 4.0
* Cognitively healthy (Mini-Mental State examination ≥ 26)
* In case of taking medications for Multiple Sclerosis: stable dosage for at least 6 months.

EXCLUSION CRITERIA:

For both healthy participants and patients:

* Contraindications to magnetic resonance imaging (metal implant in body, known claustrophobia, pacemakers)
* Severe comorbidities
* Antibiotics treatments over the last 3 months

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The groups will be selected from local community sample, hospital and general practitioners (gp).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Brain structural and functional properties | Day 1
  Brain structural and functional properties will be derived from a multi-modal Magnetic Resonance Imaging protocol.
Microbiome profile | Day 1
  Microbiome profile will be derived from a stool sample obtained from participants.

SECONDARY OUTCOMES:
Cognitive functioning | Day 1
  Cognitive functions will be measured using a neuropsychological protocol.
Concentration of blood inflammatory markers | Day 1
  A panel of key inflammatory mediators (for example, IFNgamma, IL-6, TNFalpha, IL1beta, IL10) will be evaluated in terms RNA expression level in plasma samples obtained from participants.
Eating habits | Day 1
  Information on eating habits will be derived from food questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Filippini, Principal Investigator — IRCCS San Camillo, Venezia, Italy
Locations (3):
- Italy (3):
  - IRCCS San Camillo, Venice-Lido, Venice
  - IRCCS Istituto Centro San Giovanni di Dio Fatebenefratelli, Brescia
  - Università Ca' Foscari Venezia, Venice